CLINICAL TRIAL: NCT01154751
Title: Supera Treatment Registry Observing Neointimal Growth
Brief Title: Data Registry Following Patients Using Supera Stent in the Femoral Arteries
Acronym: STRONG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment,increased loss to follow-ups and general lack of interest.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDEV Technologies, Inc.
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Peripheral Artery Disease; Femoropopliteal Artery Stenosis; Peripheral Vascular Disease
Keywords: Femoral artery stenosis; Peripheral vascular Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device SUPERA Stent (Other): SUPERA Interwoven Self-Expanding Nitinol Stent System
  Interventions: Device: SUPERA Interwoven self-expanding nitinol stent

INTERVENTIONS:
Device: SUPERA Interwoven self-expanding nitinol stent — Insertion of stent at stenotic area

SUMMARY:
Long-term, observational, prospective, multicenter registry following patients who have been implanted with the SUPERA Interwoven Self-Expanding Nitinol Stent for treating stenosis in the superficial femoral and/or femoropopliteal arteries.

DETAILED DESCRIPTION:
This registry follows up to 200 patients for at least 5 years.

The STRONG Data Registry will follow patients under real world conditions, evaluating restenosis rates, periprocedural/postprocedural complications, patency, target lesion revascularization, walking distance, stent fractures, and adverse events/serious adverse events.

ELIGIBILITY:
Exclusion Criteria:

(Clinical)

* Patient or legal guardian understands registry procedures and has voluntarily signed an informed consent in accordance with institutional and local regulatory policies. (Note: Retrospective data may be collected and entered into the EDC system after a fully executed informed consent has been provided).
* Rutherford-Becker classification 2 through 5 only
* Patient is at least 18 years of age and of legal age of consent.
* Patient must be willing to participate in the registry for at least 5 years.

(Angiographic)

* Target lesion is a single de novo or restenotic (outside a stent) SFA or Popliteal artery lesion ≥ 1 cm from origin of another stent; additional lesions may be present., but there is only one target lesion
* All SFA target lesions are to be located with the proximal point at least 2 cm below the origin of the profunda femoris artery.
* All Popliteal Artery target lesions are to be located with the most distal point at least 1 cm proximal to the bifurcation of the anterior tibial artery and the tibioperoneal trunk.
* Target lesion length 1-20 cm (visual estimate)
* Target lesion stenosis ≥50% (visual estimate)
* Popliteal artery patent if the lesion is in the SFA
* SFA patent if the lesion is in the popliteal artery
* At least one widely patent (< 50% stenosis) infrapopliteal artery (for distal run-off)

Exclusion Criteria:

(Clinical)

* Evidence of heparin induced thrombocytopenia (HIT), or intravenous tPA, Plavix, Ticlid, or aspirin therapy sensitivities
* Patient is participating in a clinical study that could confound results
* Patient is pregnant/breastfeeding at time enrollment or plans to become pregnant during the course of participation in the registry.

(Angiographic)

* Target lesion length > 20 cm
* Instent restenotic / reoccluded target lesion
* Acute (≤ 4 weeks) thrombotic occlusion
* Untreated ipsilateral pelvic stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, Prof Dr med, Principal Investigator — Herzzentrum Abteilung fur Angiologie, Bad Krozingen, Germany
Locations (4):
- Germany (4):
  - Herzzentrum Abteilung fur Angiologie, Bad Krozingen
  - Heart Center Leipzig/Park Hospital, Leipzig
  - Kathlisches Klinikum Mainz, Mainz
  - Zentrum fur Diabetes-und GefaBerkrankungen, Münster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study planned to recruit up to 200 patients across 5-10 sites in the European Union. However, during the course of the study, intake was halted at 109 patients and the registry was terminated early because of slow enrollment, increased loss to follow-ups, and general lack of interest.
Period: 6-month Follow-up
Arm/Group | Device SUPERA Stent
Started | 109
Completed | 98
Not Completed | 11
Period: 1-year Follow-up
Arm/Group | Device SUPERA Stent
Started | 98
Completed | 93
Not Completed | 5
Period: 2-year Follow-up
Arm/Group | Device SUPERA Stent
Started | 93
Completed | 83
Not Completed | 10
Period: 3-year Follow-up
Arm/Group | Device SUPERA Stent
Started | 83
Completed | 34
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 73
Region of Enrollment [Number; unit: participants]
  Germany | 109
Lesion length [Mean (Standard Deviation); unit: Centimeters] — Lesion length is site reported
  Centimeters
    Superficial femoral (n=86) | 16.40 (28.93)
    Popliteal (n=22) | 7.77 (5.00)
    Femoropopliteal conjunction (n=3) | 18.67 (2.31)
Percent diameter stenosis [Mean (Standard Deviation); unit: percentage diameter stenosis] — Percent diameter stenosis is site reported.
  percentage diameter stenosis
    Superficial femoral (n=87) | 93.07 (8.78)
    Popliteal (n=23) | 93.83 (7.91)
    Femoropopliteal conjunction (n=3) | 96.67 (5.77)
Occlusion [Number; unit: participants] — Core laboratory reported
  participants | 50

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walking Distance
Description: The Six-minute Walking Distance test is an objective method for estimation of walking capacity in patients with Peripheral Arterial Disease (PAD) or claudication.
Time Frame: At baseline
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 37
Meters | 171.30 (85.93)

2. Primary Outcome: Six-minute Walking Distance
Description: as for outcome 1
Time Frame: 30 days
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 81
Meters | 251.77 (119.44)

3. Primary Outcome: Six-minute Walking Distance
Description: as for outcome 1
Time Frame: 6 months
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 81
Meters | 263.74 (152.95)

4. Primary Outcome: Six-minute Walking Distance
Description: as for outcome 1
Time Frame: 1 Year
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 83
Meters | 262.19 (141.13)

5. Secondary Outcome: Number of Participants Experiencing Peri-procedural and Post-procedural Complications
Description: Periprocedural/Postprocedural Complications defined as complications during the procedure through 30 days post implant that include hematoma, arteriovenous (AV) fistula pseudoaneurysm, subacute occlusion, non-target lesion Percutaneous Transluminal Angioplasty (PTA) /stenting, distal embolization, and vessel perforation.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 109
Participants
  At least one | 3
  AV fistula / pseudoaneurysm | 2
  Subacute occlusion | 2
  Hematoma | 1

6. Secondary Outcome: Number of Peri-procedural and Post-procedural Complications
Description: as for outcome 5
Time Frame: 30 days
Measure: Number; unit: Number of compilcations
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 109
Number of compilcations
  At least one | 5
  AV fistula / pseudoaneurysm | 2
  Subacute occlusion | 2
  Hematoma | 1

7. Secondary Outcome: Rutherford-Becker Clinical Category
Description: Rutherford/Becker Categories:
  0 - Asymptomatic, no hemodynamically significant occlusive disease.
  1. - Mild claudication.
  2. - Moderate claudication.
  3. - Severe claudication.
  4. - Ischemic rest pain.
  5. - Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia.
  6. - Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable.
Time Frame: 30 days
Population: The number of patients analyzed is based on the data available.
Measure: Number; unit: percentage of participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 96
percentage of participants
  0 = Asymptomatic | 41.7
  1 = Mild claudication | 19.8
  2 = Moderate claudication | 18.8
  3 = Severe claudication | 13.5
  4 = Ischemic rest pain | 0.0
  5 = Minor tissue loss | 5.2
  6 = Ulceration or gangrene | 1.0

8. Secondary Outcome: Restenosis by Duplex Ultrasound
Description: In-Stent Restenosis is re-narrowing within the margins of the stent following the reduction of a previous narrowing. It is defined as the presence of a hemodynamically significant restenosis (≥ 50%), as determined by duplex ultrasonography (DUS) or arteriography. A peak systolic velocity ratio (PSVR) of 2.4 and 2.5 will be used to calculate duplex restenosis.
Time Frame: 6 months
Population: If no PSVR measurement was available, patient was excluded from restenosis analysis. If patient had TLR prior to duplex ultrasound, PSVR was excluded from restenosis analysis.
  The number of patients analyzed is based on the data available.
Measure: Number; unit: percentage of participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 91
percentage of participants
  PSVR ≥ 2.4 | 11.0
  PSVR ≥ 2.5 | 9.9

9. Secondary Outcome: Restenosis by Duplex Ultrasound
Description: as for outcome 8
Time Frame: 1 Year
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 82
percentage of participants
  PSVR ≥ 2.4 | 23.2
  PSVR ≥ 2.5 | 19.5

10. Secondary Outcome: Target Lesion Revascularization
Description: Target Lesion Revascularization (TLR): Any revascularization at the target lesion with or without evidence of target lesion diameter stenosis ≥ 50% determined by DUS or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion).
Time Frame: 6 months
Population: The number of patients analyzed is based on the data available.
Measure: Number; unit: percentage of participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 98
percentage of participants | 4.1

11. Secondary Outcome: Target Lesion Revascularization
Description: Target Vessel: The entire vessel in which the treated lesion is located. The boundaries for the iliac artery are the abdominal aortic bifurcation and the superior border of the inguinal ligament.
  Target Lesion Revascularization (TLR): Any revascularization at the target lesion with or without evidence of target lesion diameter stenosis ≥ 50% determined by DUS or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion.)
Time Frame: 1 Year
Population: The number of patients analyzed is based on the data available.
Measure: Number; unit: percentage of participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 93
percentage of participants | 11.8

12. Secondary Outcome: Stent Fracture
Description: Stent fractures determined by fluoroscopy .
Time Frame: 1 Year
Population: The number of patients analyzed is based on the data available.
Measure: Number; unit: participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 88
participants | 2

13. Secondary Outcome: Stent Fracture
Description: Stent fracture and Involuntary stent migration are types of device System Failure.
  Device System Failure is defined as the inability of the device to provide the intended clinical utility requiring surgical intervention to correct.
Time Frame: 1 to 2 years
Population: The number of patients analyzed is based on the data available.
Measure: Number; unit: participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 81
participants | 0

14. Secondary Outcome: Stent Fracture
Description: as for outcome 13
Time Frame: 1 to 3 Years
Population: The number of patients analyzed is based on the data available.
Measure: Number; unit: participants
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 33
participants | 0

15. Secondary Outcome: Target Limb Ankle Brachial Index (at Rest)
Description: Ankle Brachial Index (ABI) is a measure of the fall in blood pressure in the arteries supplying the legs and is used to detect evidence of blockages in the peripheral vessels. It is calculated by dividing the higher systolic blood pressure in the ankle (dorsalis pedis or posterior tibial) of the one leg by the higher of the two systolic blood pressures in the arms. A doppler probe is used to monitor the pulse while a sphygmomanometer is inflated above the artery. The cuff is deflated and the pressure at which the pulse returns is recorded.
  ABI=Highest Ankle Systolic Pressure/Highest Brachial Systolic Pressure
  The ABI is the ratio of the ankle to arm pressure, and an ABI between 0.9 and 1.3 is considered normal. A reduced ABI (less than 0.9) is consistent with peripheral artery occlusive disease, with values below 0.8 indicating moderate disease and below 0.5 severe disease.
Time Frame: At baseline
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 88
Ratio | 0.63 (0.29)

16. Secondary Outcome: Target Limb Ankle Brachial Index (at Rest)
Description: as for outcome 15
Time Frame: 30 days
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 84
Ratio | 1.04 (0.25)

17. Secondary Outcome: Target Limb Ankle Brachial Index (at Rest)
Description: as for outcome 15
Time Frame: 6 months
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 87
Ratio | 0.98 (0.28)

18. Secondary Outcome: Target Limb Ankle Brachial Index (at Rest)
Description: as for outcome 15
Time Frame: 1 Year
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 80
Ratio | 0.90 (0.29)

19. Secondary Outcome: Target Limb Ankle Brachial Index (at Rest)
Description: as for outcome 15
Time Frame: 2 Years
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 70
Ratio | 0.91 (0.22)

20. Secondary Outcome: Six-minute Walking Distance
Description: as for outcome 1
Time Frame: 2 Years
Population: The number of patients analyzed is based on the data available.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Device SUPERA Stent
Number analyzed (Participants) | 73
Meters | 272.75 (152.80)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Device SUPERA Stent
Serious Adverse Events (participants affected / at risk) | 84/109
Other Adverse Events (participants affected / at risk) | 87/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device SUPERA Stent (N=109)
Hospital readmittance (General disorders) | 19 (28) — Hospital Readmittance: Device-related readmittance to a care facility for a continuous period of 3 days.
Death (General disorders) | 14 (14) — Death: All-cause mortality.
Amputation (General disorders) | 2 (2) — Amputation: All-cause limb amputation.
Bleeding (Blood and lymphatic system disorders) | 1 (2) — After the perioperative period, an episode of internal or external bleeding that causes death, hospitalization, and permanent injury or necessitates transfusion of >20 cc/kg of body weight packed red blood cells in a 24-h period.
Other (General disorders) | 78 (178)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device SUPERA Stent (N=109)
Hospital readmittance (General disorders) | 19 (28) — Hospital Readmittance: Device-related readmittance to a care facility for a continuous period of 3 days.
Death (General disorders) | 14 (14) — Death: All-cause mortality.
Other (General disorders) | 81 (206)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days